CLINICAL TRIAL: NCT02557503
Title: An Randomized and Controlled Study of Hepatic Arterial Infusion of Oxaliplatin and Fluorouracil Treatment of Advanced Primary Liver Cancer After TACE
Brief Title: Hepatic Arterial Infusion of Oxaliplatin and Fluorouracil Treatment of Advanced Primary Liver Cancer After TACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Xu (Other)
Responsible Party: Sponsor-Investigator, Zhu Xu, Interventional Therapy Department, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014KT71
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-07

CONDITIONS: Advanced Adult Primary Liver Cancer
Keywords: TACE; oxaliplatin; fluorouracil; liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxaliplatin by HAIC after TACE (Experimental): To investigate the therapy effect and security of oxaliplatin on with or without concomitant vascular invasion and extrahepatic metastases unresectable advanced primary liver cancer
  Interventions: Drug: Oxaliplatin and fluorouracil
- Fluorouracil by HAIC after TACE (No Intervention): To investigate the therapy effect and security of fluorouracil on with or without concomitant vascular invasion and extrahepatic metastases unresectable advanced primary liver cancer

INTERVENTIONS:
Drug: Oxaliplatin and fluorouracil — Oxaliplatin and fluorouracil by HAIC on with or without concomitant vascular invasion and extrahepatic metastases unresectable advanced primary liver cancer after TACE
  Arms: Oxaliplatin by HAIC after TACE

SUMMARY:
To investigate the therapy effect and security of oxaliplatin and fluorouracil on with or without concomitant vascular invasion and extrahepatic metastases unresectable advanced primary liver cancer

ELIGIBILITY:
Inclusion Criteria:

1. With written informed consent
2. Age ranged from 18 to 80 years, both men and women
3. Confirmed by pathology or clinical diagnosis of liver cancer
4. Progress systemic chemotherapy or who can not tolerate chemotherapy, or who refuse chemotherapy
5. Never received TACE treatment
6. (M) RECIST 1.0 criteria measurable liver lesions at several ≥2, each lesion diameter ≥3 cm long and ≤20cm,
7. ECOG PS score of ≤2
8. expected survival time ≥12 weeks
9. The test results before 7 days entered the group must meet the following requirements:

Hemoglobin ≥ 90 g / L Absolute neutrophil count (ANC)> 1,500 / mm3 Platelet count ≥ 80x109 / L Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5 times the upper limit of normal (UNL) Total bilirubin <3UNL Serum creatinine <1.5 UNL PT or INR, PPT <1.5 UNL (for patients undergoing warfarin or heparin anticoagulant therapy, if there is no evidence that there is an abnormality of the above parameters, you can enter the group, but must be closely monitored to detect at least once a week until the INR stable)

Exclusion Criteria:

1. Specific circumstances of patients not suitable for TACE therapy / chemotherapy
2. Hepatic decompensation, or the presence of hepatic encephalopathy
3. Before entering the study with gastrointestinal bleeding within 30 days
4. Presence of brain metastasis
5. Pregnant or lactating women
6. Active bleeding or sepsis
7. History of heart disease:

   NYHA two or more of congestive heart failure, symptomatic coronary artery disease Need to use β-blockers or digoxin medication other than arrhythmias
8. Despite treatment, still systolic blood pressure> 150 mmHg or diastolic blood pressure> 90 mmHg hypertension
9. Not cure severe trauma, acute or incurable ulcer, or three months fracture
10. The researchers believe their poor compliance
11. Exist once or primary lesion or histologically different tumors and colorectal cancer, except: head and neck carcinoma in situ, cured basal cell carcinoma, superficial bladder cancer (Ta, Tis, T1), and the group 3 years ago, it has been cured of cancer
12. HIV infection or the presence of AIDS-related illness, or severe acute and chronic diseases
13. Drug abuse, or suffering that could interfere with study compliance and other psychological or psychiatric disorders
14. Need drug therapy epilepsy (such as steroids or antiepileptic drugs
15. Chemotherapy contraindications exist
16. Any instability or likely to endanger the patient in this study the safety and compliance of the case

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | three years

SECONDARY OUTCOMES:
overall survival (OS) | three years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China